CLINICAL TRIAL: NCT04074304
Title: Developing and Piloting a Multi-component Technology-based Care Intervention to Address Patient Symptoms and Caregiver Burden in Home Hospice
Brief Title: Developing and Piloting a Multi-component Technology-based Care Intervention to Address Patient Symptoms and Caregiver Burden in Home Hospice. Phase 1.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Visiting Nurse Service of New York (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-11022933 frmrly 19-04020138; 1K76AG059997-01A1 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-03

CONDITIONS: Home Hospice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I-HoME prototype (Other): Participants will be shown prototype of I-HoME and provide feedback as part of the user-center design process.
  Interventions: Other: I-HoME

INTERVENTIONS:
Other: I-HoME — A multi-component technology-based care intervention.

SUMMARY:
With the growth of hospice, older adults have the opportunity to receive home-based care aimed at reducing suffering and focusing on quality of life at the end of life. While use of technology and educational videos has yet to be fully developed, structured, and evaluated in home hospice care, it has shown promise to improve care in other settings. Therefore, this study aims to develop and evaluate a multi-component technology-based care intervention, i.e., Improving Home hospice Management of End of life issues through technology (I-HoME), that focuses on assessing and addressing patient symptoms and caregiver burden in the home hospice setting through synchronous live video visits and educational videos. The aim of the first phase of the project is to employ an iterative user-centered design process to develop I-HoME for home hospice patients and their caregivers prior to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Home hospice providers (N=10) and family caregivers (N=10) must be English speaking, 18 years of age or older, not blind, and either providing or receiving home hospice care. Home hospice patients (N=10) must be English speaking, 65 years of age or older, not blind, and enrolled in home hospice care.

Exclusion Criteria:

* Patients with a terminal diagnosis of dementia or patients who have cognitive impairment and unable to sign a written informed consent will be excluded.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Participants' experience using the intervention as measured by the I-HoME User-centered design questionnaire | 1 day
  A questionnaire consisting of open ended questions asking participants to provide feedback and their thoughts about the I-HoME intervention. The responses gathered are not scored, but qualitative analysis will be performed to identify issues that will be used to make revisions to the I-HoME intervention before starting phase 2 of the project.

CONTACTS AND LOCATIONS:
Overall Officials: Veerawat Phongtankuel, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The Visiting Nurse Service of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No